CLINICAL TRIAL: NCT06110429
Title: Sodium Lactate Versus Hypertonic Saline Solution in the Treatment of Intracranial Hypertensive Episodes in Severe Brain Injured Patients
Acronym: SLHYSS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Hervé Quintard, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 701546
Record Dates: First submitted 2023-04-18; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Intra Cerebral Hypertension; Lactate Sodium Solution
Keywords: intracerebral hypertension; lactate sodium
MeSH Terms: interventions — Sodium Lactate; Saline Solution, Hypertonic

STUDY DESIGN:
Intervention Model Description: A prospective open randomized single center study comparing Sodium lactate (SL) to Hypertonic Saline Solution (HSS) in brain injured adult ICU
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lactate sodium (Experimental): 100 mL of Sodium lactate (Osmolality 2560 mOsm/L) in 15 mins of administration via a central venous catheter
  Interventions: Drug: Lactate, Sodium
- Hypertonic Saline solution (Active Comparator): single infusion of 100 mL of 7.5% saline (osmolarity, 2560 mOsm/L) (HSS group)in 15 mins of administration via a central venous catheter
  Interventions: Drug: Hypertonic saline

INTERVENTIONS:
Drug: Lactate, Sodium — Isovolemic and osmotic infusion Comparison of osmotic agent
  Arms: lactate sodium
Drug: Hypertonic saline — Isovolemic and osmotic infusion Comparison of osmotic agent
  Arms: Hypertonic Saline solution

SUMMARY:
Brain oedema is a major complication of brain injury (TBI). It increases the risk of intracranial hypertension (ICH) and brain hypoxia, leading to an increase in mortality and poor neurologic outcome. Increased water content in the injured brain can be related to a vasogenic or cellular pathway. Osmotherapy, by using mannitol or hypertonic saline (HSS), is recommended and currently administered for the treatment of ICH in this setting. Beside these two usual treatments, sodium lactate (SL), a metabolic and neuroprotective solution, has recently been described as having similar effects on lowering intracranial pressure (ICP). In a previous study, conducted in patients with severe TBI, (1) Ichai et al. reported that a bolus of half-molar SL was as effective than equimolar doses of mannitol to reduce elevated ICP (less refractory ICH and higher and longer reduction of ICH).

Objective(s):

The purpose of the study is to analyze the effect on ICH of SL compared to a hypertonic saline solution (HSS).

Outcome(s):

The primary endpoint is the efficacy in lowering ICH after 4 h. Secondary endpoints were percentage of successfully treated episodes of intracranial hypertension and neurological status at discharge from ICU.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an acute, isolated, severe brain injury (SAH, TBI, ICH)
* Glasgow coma score <8
* Monitored using ICP device
* Presenting an episode of intracranial hypertension requiring osmotherapy. ( defined as increase in ICP 25 mmHg which persisted for more than 5 min in the absence of noxious stimulations)
* Informed Consent as documented by signature

Exclusion criteria

* Pregnant woman
* Bilateral fixed dilatated pupils
* Initial hypernatremia (>155 mmol/l)
* Penetrating head injury
* Active participation to another trial (Clin B, C)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
intracranial pressure (ICP) | 240 minutes
  Invasive monitoring of intracranial pressure

SECONDARY OUTCOMES:
Percentage of successfully treated episodes | 48 hours
  decrease of ICP >5mmHg or level <20mmHg
Oxygen tissular pressure | 240 minutes
  In vasive measurement of tissular pressure
Neurological status at discharge of ICU | through study completion, an average of 30 days
  Measurement Glasgow Outcome Scale
Number of episodes of intracranial hypertension | through study completion, an average of 30 days
  Number of episodes of intracranial hypertension

IPD SHARING:
Plan to Share IPD: No